CLINICAL TRIAL: NCT03423966
Title: Effect of the Use of Smartphone Pedometers on the Weight of Overweight and Obese Clients at the General Outpatient Department, National Hospital Abuja.
Brief Title: Smartphone Pedometers and Body Mass of Overweight and Obese Clients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Hospital, Abuja (Other Government)
Responsible Party: Principal Investigator, Ngong Hipoletus Cyprian, Senior Registrar and Secretary, Research and Academic Committee, National Hospital, Abuja
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHA/EC/088/2017
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Objective Mobility Evaluation (Experimental): Usual Care Plus a Smartphone pedometer App
  Interventions: Device: Smartphone Pedometer App
- Usual Care (UC) (No Intervention): Usual Care of obesity

INTERVENTIONS:
Device: Smartphone Pedometer App — Installation of the free pedometer app and explanation to participants to target 10000 steps per day. The intent is not the accuracy of the pedometer but the motivation especially to a community yet to harness the full potentials of the mobile phone technology
  Arms: Self Objective Mobility Evaluation

SUMMARY:
The study sets out to determine the effect of smartphone pedometers on the body mass of overweight and obese clients at the general outpatient department, national hospital Abuja.

It is a synopsis of the proposed dissertation submitted to the West African College of Physicians in partial fulfillment of the requirements for the part 11 Fellowship examination of the faculty of Family Medicine.

DETAILED DESCRIPTION:
3.1 Study Area The Hospital is a melting pot of referral cases, fresh cases, executive patients and the masses alike and therefore gives a scout picture of the non-communicable diseases situation in Nigeria. First contact to undifferentiated patients is offered in the clinic. It is accredited by both the West African College of Physician and the National Postgraduate Medical College of Nigeria for residency training in Family Medicine.

3.2 Study Population The study will be carried out among consenting adult overweight and obese patients attending the GOPC of National Hospital Abuja.

3.3 Study Design This study is a Randomized Controlled Trial with parallel open label design.

3.4 Duration of Study The study will be conducted over a period of 24 weeks with a lead in period of 4 weeks for recruitment.

3.5 Minimum Sample Size Estimation The minimum sample size was calculated using the formula for sample size estimation for tests between two independent means.

N = 2 s 2 (zcrit+ zpower)2 D2 Where N = Sample size estimate zcrit = critical value for alpha (0.05 alpha has a zcrit of 1.960 zpower = value for 1-beta (80% power has a z of 0.842) s = standard deviation D = the expected difference between the two means (i.e. the minimum difference between the two means that will be considered clinically significant).

From a previous study that considered weight loss as the primary outcome in black women, the standard deviation was 3.479 A difference in means of 1.44 kg is regarded as clinically significant. Therefore, the sample size calculated for the weight variable in each arm of the investigation will be; N = 2×3.42 (1.960+ 0.842)2/ 1.44 squared = 87.5 for each arm of the study and a total of 176 participants.

The minimum sample size for the study is therefore 176. Being a medium term duration study, we assume a maximum attrition rate of 10%, the final sample size to recruit is 194, with 97 participants in each arm of the study.

3.7 Study Instruments and Tools The data capture form broadly consists of 6 sections and incorporates the fundamental aspects of an obesity consultation clinic; Android phone versions higher than 3.0 with a Pedometer app version 5.19 by tayutau which is a simple easy to use pedometer application that measures steps for physical activity monitoring. It has three modes that count the steps, the distance or the calories burnt. It has the advantage of recording at least 2 months of daily step counts and can be evaluated at leisure in the clinic. It also shows your average pace.

Stadiometer: (By SECA; Vogel and Halke; made in Germany) will be used for height measurements (cm).

Weighing Scale: (By SECA; Vogel and Halke; Made in Germany) will be used for weight measurements (kg).

Sphygmomanometer: (Dekamet Accoson Mercury Sphygmomanometer, Made in England). Calibrated in mmHg from 0 - 300 mmHg; arm cuff size 22 - 32(cm); will be used for blood pressure measurements (mmHg).

Tape rule measure: Flexible, non-stretchable tape measure (NEWEY, Made in Germany). Calibrated in (cm), from 0 - 150, will be used for WC measurements.

3.8 Study Procedure 3.81 Research Assistants Four research assistants will be trained in the research proceedings including the initial screening, inclusion and exclusion criteria. The research assistants are also resident doctors who have basic experience in the management of obese clients.

3.82 Screening for Eligibility Screening for eligibility will be conducted at the first visit in the General Outpatient Clinic by 4 trained research assistants. The age of the prospective participant, ownership of a pedometer capable phone, the Body Mass Index and a pass in the Physical Activity Readiness Questionnaire (PARQ) will be the minimum to proceed to the randomization and study clinic.

A "Yes" response to any question in the PARQ requires further evaluation and depending on severity, may render a participant ineligible for participation.

3.83 Randomization and Allocation Concealment At the study clinic, eligible consenting participants will be randomized to the two arms of the study. Allocation concealment will be achieved by using opaque envelopes containing allocation color coded cards, white for 'UC' and pink for 'SOME' will be used to execute random assignment to the two group. Under supervision of a research assistant, participants will pick one of the envelopes before proceeding to the consulting room without opening the envelope for enrollment. Allocation ratio will be 1:1.

Randomization will be achieved by having prospective participants pick color coded cards before anthropometric examinations. After every pick, the envelopes will be reshuffled before the next pick. The color coded cards will be stuck on the front inner cover of folders of all participants to avoid confusion. They will be no formal blinding.

3.84 Aspects Common to Both Study Arms After signing the consent form, all eligible participants will fill out a brief health-screening and qualification questionnaire within the data capture form. Participants will all have the International Physical Activity Questionnaire Short Form (IPAQ-SF) tools computed at the beginning to assess the level of physical activity, at 8 weeks and at the end of the study (16 weeks) with results computed into a continuous variable by the formula; Total MET/Min/week = [Walking METs × min × days] + [Moderate METs × min × days] + [Vigorous METs × min × days] and finally grouped into categorical variables of low, moderate and high physical activity levels.

Participants will be counseled using the 5A model and given an exercise prescription to maintain for the duration of the study. They will be counseled on dietary modifications and exercise plans. Basic lifestyle counseling will be in the form of a uniform lifestyle "SERVE" advice slip modified from the one used by the Montefiore Medical Center, Albert Einstein College of Medicine and New York University School of Medicine as reported by Sheira Schlair, Sarah Moore, Michelle McMacken, and Melanie Jay for both groups with the printed leaflets given to participants.

Participants will be offered the routine care of their presenting complaint. Blood pressure will be measured at the beginning, at 8 weeks and at 16 week using an Omron blood pressure with appropriate cuffs. Baseline assessment will include anthropometric measurements - height (measured in bare feet to nearest 0.5 cm using a stadiometer) at the beginning of the study only, weight (measured to nearest 0.1 kg), waist and neck circumferences will be measured using a flexible measuring tape between the middle of the bottom rib (close to the navel) and iliac crest and recorded to the nearest 0.1 cm. These measurements will be taken at the beginning, at 8 weeks and at the end of the 16 weeks. Participants' phone numbers will be collated for bulk text message reminders of exercise prescription.

3.85 Aspects only Common to Intervention Group Only At this juncture, the balloted envelop will be opened and if participants belong to the SOME group, they will now have the Pedometer app installed on their smartphones and calibrated with a 100 step test for sensitivity. They will be shown how to use the application and instructed to keep their phones handy, charged and chart their step count and monitor the increment. They will be a step count record card with targets in slow increments to 10,000 steps per day.

3.86 Retention Efforts

Retention will be promoted by:

1. Examining and attempting to remove barriers (e.g., adjusting clinic hours)
2. Positive attitude and demeanor towards overweight and obesity with investigators training in motivational methods and the sensitivity of obesity lingua. (Use "weight problem" instead of "obesity")
3. Give incentives such as educational materials and web links to keep participants active and give them ownership of the problem. They will also be an incentivizing prize for the best 5 completers of the trial in terms of weight outcome.
4. The trial will make every effort to maintain contact with inactive participants via phone, e-mail and text messaging to continue encouraging participants.

3.87 Follow up, Monitoring and Evaluation They shall be at least two follow ups per participant during which further evaluations and weight measurement of primary and secondary outcomes will be conducted. For comorbidities that require more frequent follow up, this will be pursued to a logical conclusion.

3.9 Data Collection A pretested investigator administered data capture form will be used to collect demographic data and baseline anthropometric and laboratory evaluation will be conducted. participants will be given appropriate care and follow up. A further set of evaluation will be obtained at 8 weeks and the end of the study.

4.1 Ethical Consideration Approval to conduct the study has been obtained from the Research Ethics Committee of the National Hospital, Abuja and the study shall be conducted based on good clinical practice principles and in conformity with the Declaration of Helsinki.

Written informed consent shall be obtained from each participant. No participant will be coerced. Welfare, rights and confidentiality shall be guaranteed for all participants. Only serial numbers will be allocated to participants and their names will not be entered into the data capture forms. However, phone numbers will be required for adequate follow up.

Consultations and physical examination will be done in privacy with participants' caregiver or a chaperone in attendance during physical examination. Undue discomfort will be avoided. The issues of weight will be discussed in a sensitive manner and local cultures will be respected during the study.

4.2 Data Analysis Data will be collected and collated in Microsoft Excel spreadsheet from Windows Office Package Version 8. Data will then be exported and analyses will be conducted using Statistical Package for the Social Sciences version 20.0 for Windows software with a p value of <0.05 used to indicate statistically significant differences (V.20.0, 2010; SPSS, Inc., Chicago, Illinois, USA). The data will be analyzed for normality and descriptively. Data transformation will be conducted on data that are not normally distributed.

Descriptive statistics such as the mode, median, mean and standard deviation will be used to analyze all demographic data and primary and secondary outcome variables. Independent t-tests (for continuous data) and chi-square tests (for categorical data) will be used to compare at baseline, the demographic and outcome variables between the two groups.

Two-way repeated-measures analysis of covariance will be conducted to compare the effects of using a pedometer on the primary outcome measure. The intention-to-treat principle (last observation carried forward) will be used to handle missing data resulting from dropout. In addition, an independent t-test will be used to compare the average physical activity level between the two groups.

4.4 Budget

1. Investigator's Assistants for data collection (x 4 assistants) 30,000.00 x 5= N150,000.00
2. Fasting Blood Glucose investigation (at N400 per participant); N400 x 125= N50,000.00
3. Data for installation ( at N9,000.00 per month) N9,000.00 x 4 = N36,000.00
4. Photocopy of Study Materials (i.e. consent form, case report form, etc) = 100,000.00 GRAND TOTAL 340,000.00 NGA

ELIGIBILITY:
Inclusion Criteria:

1. Consenting screened participants that are overweight or obese who want to lose at least 5% of their baseline weight.
2. Adults aged 18 to 65 years old.

Exclusion Criteria:

1. Clients on weight lose drugs because this may confound the cause of the weight loss.
2. Patients with conditions that do not allow mobility.
3. Patients with major organ failure because such patients may not be so stable to cope with prescribed exercise schedule.
4. Pregnancy; present, intending and 6 months postpartum because the cause of the weight loss or gain may be attributed to the pregnancy.
5. Morbidly obese clients because this are candidates for drug therapy and surgical interventions and it will be unethical to delay such interventions.
6. Clients with no android smartphone that are randomized to the intervention group because the intervention will not be possible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 4 months
  Changes in weight after the use of pedometer app

SECONDARY OUTCOMES:
Body Mass Index | 4 month
  Changes in BMI after intervention
Waist Circumference | 4 Months
  Changes in waist circumference with intervention
Blood Pressure | 4 months
  Changes in Blood pressure with intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ngong H Cyprian, MBBS, Principal Investigator — National Hospital, Abuja
Locations (1):
- National Hospital Abuja, Abuja, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: No
I will not share the raw data